CLINICAL TRIAL: NCT03923101
Title: The Homburg Keratoconus Center (HKC) - a Keratoconus Observation Study
Brief Title: The Homburg Keratoconus Center (HKC)
Status: Recruiting | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Elias Flockerzi, Principal Investigator, Resident of Ophthalmology, University Hospital, Saarland
Other Study IDs: HKC
Record Dates: First submitted 2019-03-22; First posted 2019-04-22 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Keratoconus
Keywords: Keratoconus; Crosslinking; Intracorneal ring segments; Gas-permeable rigid contact-lenses; Penetrating Keratoplasty; Deep anterior lamellar Keratoplasty; ABCD Grading System
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Keratoconus: Aim is to include as many Keratoconus patients as possible with the intention to elucidate how the disease begins and develops during lifetime.
  Interventions: Diagnostic Test: Topographic, tomographic and biomechanical analysis.

INTERVENTIONS:
Diagnostic Test: Topographic, tomographic and biomechanical analysis. — The study is based upon data obtained during routine medical follow-ups using
  1. the Pentacam high resolution (Oculus, Wetzlar, Germany)
  2. the Corvis ST (Oculus, Wetzlar, Germany)
  3. the Anterior-Segment Optical Coherence Tomograph (AS-OCT) Casia 2 (Tomey, Nagoya, Japan)
  4. the Ocular Response Analyzer (Reichert Technologies, New York, USA).

SUMMARY:
Aim of this study is to conduct longitudinal and cross-sectional analyses about the corneal ectatic disease Keratoconus based on data obtained from Keratoconus patients in the Homburg Keratoconus Center (HKC).

The Homburg Keratoconus Center (HKC) was founded in 2010 and, up to now, comprises more than 3,000 Keratoconus patients. Topographic, tomographic and biomechanic characteristics of the disease are being analyzed with the intention to elucidate how the disease begins and develops during lifetime.

ELIGIBILITY:
Inclusion Criteria:

* All Keratoconus patients presenting in the department of ophthalmology, Saarland University Medical Center, Homburg, Saarland, Germany.

Exclusion Criteria:

* Patients without Keratoconus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Keratoconus patients of all ages presenting in the department of ophthalmology, Saarland University Medical Center, Homburg, Saarland, Germany, should be included.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
An overview about development of anterior corneal curvature in Keratoconus disease during lifetime. | 01/01/2011-01/01/2019
  The anterior radius of curvature (ARC, 3mm zone) of Keratoconus patients as measured by the Pentacam high resolution (Oculus, Wetzlar, Germany) at different ages (according to: Belin MW and Duncan JK. Keratoconus: The ABCD grading system. Klin Monbl Augenheilkd. 2016; 233(6): 701-707) is put into relation to the age of the Keratoconus patients.
An overview about development of posterior corneal curvature in Keratoconus disease during lifetime. | 01/01/2011-01/01/2019
  The posterior radius of curvature (PRC, 3mm zone) of Keratoconus patients as measured by the Pentacam high resolution (Oculus, Wetzlar, Germany) at different ages (according to: Belin MW and Duncan JK. Keratoconus: The ABCD grading system. Klin Monbl Augenheilkd. 2016; 233(6): 701-707) is put into relation to the age of the Keratoconus patients.
An overview about development of the thinnest corneal pachymetry in Keratoconus disease during lifetime. | 01/01/2011-01/01/2019
  The thinnest corneal pachymetry of Keratoconus patients as measured by the Pentacam high resolution (Oculus, Wetzlar, Germany) at different ages (according to: Belin MW and Duncan JK. Keratoconus: The ABCD grading system. Klin Monbl Augenheilkd. 2016; 233(6): 701-707) is put into relation to the age of the Keratoconus patients.
An overview about development of the best corrected distance visual acuity in Keratoconus disease during lifetime. | 01/01/2011-01/01/2019
  The best corrected distance visual acuity of Keratoconus patients as raised as part of the clinical examination at different ages (according to: Belin MW and Duncan JK. Keratoconus: The ABCD grading system. Klin Monbl Augenheilkd. 2016; 233(6): 701-707) is put into relation to the age of the Keratoconus patients.
Reproducibility study: Kmax. | 01/01/2011-01/01/2019
  Measurements of Kmax measured by different devices (Pentacam high resolution, Oculus, Wetzlar, Germany; Anterior-Segment Optical Coherence Tomograph (AS-OCT) Casia 2, Tomey, Nagoya, Japan) are being compared and set into relation at different Keratoconus stages with the intention to investigate, whether measurement inaccuracies occur at later Keratoconus stages using different devices.
Reproducibility study: Thinnest corneal pachymetry. | 01/01/2011-01/01/2019
  Measurements of the thinnest corneal pachymetry as measured by different devices (Pentacam high resolution, Oculus, Wetzlar, Germany; Anterior-Segment Optical Coherence Tomograph (AS-OCT) Casia 2, Tomey, Nagoya, Japan) are being compared and set into relation at different Keratoconus stages with the intention to investigate, whether measurement inaccuracies occur at later Keratoconus stages using different devices.
Reproducibility study: Thinnest corneal pachymetry at the apex position. | 01/01/2011-01/01/2019
  Measurements of the thinnest corneal pachymetry at the apex position as measured by different devices (Pentacam high resolution, Oculus, Wetzlar, Germany; Anterior-Segment Optical Coherence Tomograph (AS-OCT) Casia 2, Tomey, Nagoya, Japan) are being compared and set into relation at different Keratoconus stages with the intention to investigate, whether measurement inaccuracies occur at later Keratoconus stages using different devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flockerzi E, Seitz B. Keratectasia severity staging and progression assessment based on the biomechanical E-staging. Eye Vis (Lond). 2024 Jul 1;11(1):24. doi: 10.1186/s40662-024-00392-3. PMID 38946004
- [Background] Sideroudi H, Flockerzi E, Daas L, Jullien T, Xanthopoulou K, Hamon L, Seitz B. Baseline Characteristics of 1976 Patients With Ectatic Corneal Disorders at a Single Center From 2010 to 2021: A Cross-Sectional Study of the Homburg Keratoconus Center. Eye Contact Lens. 2023 Sep 1;49(9):392-398. doi: 10.1097/ICL.0000000000001014. Epub 2023 Jul 14. PMID 37458424
- [Background] Flockerzi E, Vinciguerra R, Belin MW, Vinciguerra P, Ambrosio R Jr, Seitz B. Combined biomechanical and tomographic keratoconus staging: Adding a biomechanical parameter to the ABCD keratoconus staging system. Acta Ophthalmol. 2022 Aug;100(5):e1135-e1142. doi: 10.1111/aos.15044. Epub 2021 Oct 16. PMID 34655452
- [Background] Flockerzi E, Elzer B, Daas L, Xanthopoulou K, Eppig T, Langenbucher A, Seitz B. The Reliability of Successive Scheimpflug Imaging and Anterior Segment Optical Coherence Tomography Measurements Decreases With Increasing Keratoconus Severity. Cornea. 2021 Nov 1;40(11):1433-1439. doi: 10.1097/ICO.0000000000002657. PMID 34633357
- [Background] Flockerzi E, Vinciguerra R, Belin MW, Vinciguerra P, Ambrosio R Jr, Seitz B. Correlation of the Corvis Biomechanical Factor with tomographic parameters in keratoconus. J Cataract Refract Surg. 2022 Feb 1;48(2):215-221. doi: 10.1097/j.jcrs.0000000000000740. PMID 34321407
- [Background] Flockerzi E, Hafner L, Xanthopoulou K, Daas L, Munteanu C, Langenbucher A, Seitz B. Reliability analysis of successive Corneal Visualization Scheimpflug Technology measurements in different keratoconus stages. Acta Ophthalmol. 2022 Feb;100(1):e83-e90. doi: 10.1111/aos.14857. Epub 2021 Mar 22. PMID 33750037
- [Background] Flockerzi E, Xanthopoulou K, Goebels SC, Zemova E, Razafimino S, Hamon L, Jullien T, Kluhspies U, Eppig T, Langenbucher A, Seitz B. Keratoconus staging by decades: a baseline ABCD classification of 1000 patients in the Homburg Keratoconus Center. Br J Ophthalmol. 2021 Aug;105(8):1069-1075. doi: 10.1136/bjophthalmol-2020-316789. Epub 2020 Aug 23. PMID 32830125
- [Derived] Flockerzi E, Xanthopoulou K, Daas L, Feld S, Langenbucher A, Seitz B. Evaluation of Dynamic Corneal Response Parameters and the Biomechanical E-Staging After Accelerated Corneal Cross-Linking in Keratoconus. Asia Pac J Ophthalmol (Phila). 2022 Nov 1;11(6):514-520. doi: 10.1097/APO.0000000000000580. PMID 36417675